CLINICAL TRIAL: NCT04500496
Title: Vaginal Dinoprostone Versus Vaginal Isonicotinic Acid Hydrazide Prior to Diagnostic Office Hysteroscopy in Postmenopausal Patients: a Randomized Controlled Trial
Brief Title: Vaginal Dinoprostone Versus Isonicotinic Acid Hydrazide Prior to Diagnostic Office Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/351/4/19
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Postmenopausal Bleeding
MeSH Terms: interventions — Isoniazid; Dinoprostone; KLK15 protein, human

STUDY DESIGN:
Intervention Model Description: open label randomized controlled study
Masking Description: open label randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 tablet of INH 900 mg inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: INH
- dinoprostone (Active Comparator): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: dinoprostone

INTERVENTIONS:
Drug: INH — 3 tablet of INH inserted by the patient 12 hours before the scheduled office hysteroscopy
  Other Names: Isonicotinic acid hydrazide
  Arms: INH
Drug: dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Other Names: prostin
  Arms: dinoprostone

SUMMARY:
To compare the effectiveness of vaginal dinoprostone and vaginal Isonicotinic acid hydrazide in minimizing the pain experienced by postmenopausal patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopist.

DETAILED DESCRIPTION:
hysteroscopy is commonly used in the diagnosis and treatment of intrauterine lesions such as polyps, ﬁbroids, septa, and adhesions, and in the presence of abnormal bleeding and during the removal of an intrauterine device or foreign body. Cervical ripening is made possible by the use of medication through different routes.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for ofﬁce hysteroscopy (postmenopausal bleeding or abnormal ultrasound ﬁndings)

Exclusion Criteria:

* Nulliparous patients
* patients with cervical pathology
* retroverted uterus (detected by transvaginal ultrasound)
* previous cervical surgery
* patients with severe vaginal bleeding
* allergy or contraindications to dinoprostone or INH therapy

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Menopausal patients with an indication for ofﬁce hysteroscopy
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 10 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure. Visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Operative time | 15 minutes
  From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination
Pain intensity will be assessed by visual analogue scale | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure. Visual analogue scale ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No